CLINICAL TRIAL: NCT03832179
Title: Steroid vs. Anti-vascular Endothelial Growth Factor for Diabetic Macular Edema Prior to Phacoemulsification
Acronym: STAMP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bay Area Retina Associates (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Caesar Luo, MD, FACS, Physician, Bay Area Retina Associates
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAMP
Record Dates: First submitted 2019-02-05; First posted 2019-02-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Macular Edema; Cataract
MeSH Terms: conditions — Cataract | interventions — Bevacizumab; Ranibizumab; aflibercept; Calcium Dobesilate; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Two parallel groups, one group receiving anti-vascular endothelial growth factor and the other group receiving Ozurdex.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Anti-vascular endothelial growth factor (Active Comparator): Intravitreal Bevacizumab, Ranibizumab, or Aflibercept
  Interventions: Drug: Bevacizumab; Drug: Ranibizumab; Drug: Aflibercept
- Ozurdex (Experimental): Intravitreal Ozurdex
  Interventions: Drug: Ozurdex

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab
  Other Names: Avastin
  Arms: Anti-vascular endothelial growth factor
Drug: Ranibizumab — Ranibizumab
  Other Names: Lucentis
  Arms: Anti-vascular endothelial growth factor
Drug: Aflibercept — Aflibercept
  Other Names: Eylea
  Arms: Anti-vascular endothelial growth factor
Drug: Ozurdex — Ozurdex
  Other Names: Dexamethasone implant
  Arms: Ozurdex

SUMMARY:
The primary objective of this study is to compare the efficacy of antecedent intravitreal anti-vascular endothelial growth factor therapy vs. Ozurdex in reducing post-cataract surgery related macular edema in patients with pre-existing diabetic macular edema.

DETAILED DESCRIPTION:
In patients with pre-existing diabetic macular edema, anti-vascular endothelial growth factor therapy (Bevacizumab, ranibizumab, or aflibercept) will be compared to Ozurdex therapy administered 1 week prior to phacoemulsification cataract extraction. Spectral domain optical coherence tomography and visual acuity will be acquired at 1 week, 1 month, 2 months, and 3 months following cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of age
* Gender- All
* Race- All
* Diagnosis of Diabetes (Type 1 or 2) with a concomitant diagnosis of diabetic macular edema as demonstrated on spectral domain optical coherence tomography (Heidelberg Spectralis)
* >250 microns central foveal thickness
* Able and willing to provide informed consent

Exclusion Criteria:

* Significant renal disease
* A condition that in the opinion of the investigator would preclude participation
* Participation in another investigational trial within 30 days of randomization
* Application of focal macular laser within 120 days of enrollment
* Administration of Iluvien implant within 3 years of enrollment
* Administration of intravitreal triamcinolone within 3 months of enrollment
* Administration of any anti-vascular endothelial growth factor agent within 30 days of enrollment
* Known hypersensitivity to any of the investigational products
* Blood pressure >180/110
* Women who are pregnant, lactating, or intend to become pregnant within 1 year of randomization
* Vulnerable populations- including but not limited to wards of the state, cognitively impaired individuals, prisoners, institutionalized individuals
* Individual is planning on moving within 6 months of study enrollment
* Macular edema secondary to cause other than diabetic macular edema
* Ocular condition that, in the opinion of the investigators, may affect course of macular edema during course of study (vein occlusion, uveitis, etc.)
* Evidence of ocular infections
* Evidence of uncontrolled glaucoma
* Known hypersensitivity to any components of bevacizumab, ranibizumab, aflibercept, or Ozurdex

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Comparison of central foveal thickness outcomes of anti-vascular endothelial growth factor vs. Ozurdex therapy | 3 months after cataract surgery
  Central foveal thickness will be measured in microns by spectral domain optical coherence tomography (Heidelberg) and compared to baseline at post-operative week 1, postoperative month 1, postoperative month 2, and postoperative month 3 for both anti-vascular endothelial growth factor and Ozurdex groups

SECONDARY OUTCOMES:
Visual acuity outcomes of anti-vascular endothelial growth factor vs. Ozurdex therapy | 3 months after cataract surgery
  Snellen visual acuity will be measured and converted into logMAR and compared to baseline at post-operative week 1, postoperative month 1, postoperative month 2, and postoperative month 3 for both anti-vascular endothelial growth factor and Ozurdex groups

CONTACTS AND LOCATIONS:
Overall Officials: Caesar Luo, MD, Principal Investigator — Physician
Locations (1):
- Bay Area Retina Associates, Walnut Creek, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rauen PI, Ribeiro JA, Almeida FP, Scott IU, Messias A, Jorge R. Intravitreal injection of ranibizumab during cataract surgery in patients with diabetic macular edema. Retina. 2012 Oct;32(9):1799-803. doi: 10.1097/IAE.0b013e31824bebb8. PMID 22495327
- [Background] Furino C, Boscia F, Niro A, Giancipoli E, Grassi MO, D'amico Ricci G, Blasetti F, Reibaldi M, Alessio G. Combined Phacoemulsification and Intravitreal Dexamethasone Implant (Ozurdex(R)) in Diabetic Patients with Coexisting Cataract and Diabetic Macular Edema. J Ophthalmol. 2017;2017:4896036. doi: 10.1155/2017/4896036. Epub 2017 Aug 13. PMID 28884024
- [Background] Calvo P, Ferreras A, Al Adel F, Dangboon W, Brent MH. EFFECT OF AN INTRAVITREAL DEXAMETHASONE IMPLANT ON DIABETIC MACULAR EDEMA AFTER CATARACT SURGERY. Retina. 2018 Mar;38(3):490-496. doi: 10.1097/IAE.0000000000001552. PMID 28196056
- [Background] Yumusak E, Ornek K. Comparison of Perioperative Ranibizumab Injections for Diabetic Macular Edema in Patients Undergoing Cataract Surgery. J Ophthalmol. 2016;2016:7945619. doi: 10.1155/2016/7945619. Epub 2016 Jul 14. PMID 27493795
- [Background] Lim LL, Morrison JL, Constantinou M, Rogers S, Sandhu SS, Wickremasinghe SS, Kawasaki R, Al-Qureshi S. Diabetic Macular Edema at the time of Cataract Surgery trial: a prospective, randomized clinical trial of intravitreous bevacizumab versus triamcinolone in patients with diabetic macular oedema at the time of cataract surgery - preliminary 6 month results. Clin Exp Ophthalmol. 2016 May;44(4):233-42. doi: 10.1111/ceo.12720. Epub 2016 Mar 29. PMID 26871700
- [Background] Schmier JK, Halpern MT, Covert DW, Matthews GP. Evaluation of costs for cystoid macular edema among patients after cataract surgery. Retina. 2007 Jun;27(5):621-8. doi: 10.1097/01.iae.0000249577.92800.c0. PMID 17558326
- [Background] Hayashi K, Igarashi C, Hirata A, Hayashi H. Changes in diabetic macular oedema after phacoemulsification surgery. Eye (Lond). 2009 Feb;23(2):389-96. doi: 10.1038/sj.eye.6703022. Epub 2007 Oct 26. PMID 17962820
- [Background] Hartnett ME, Tinkham N, Paynter L, Geisen P, Rosenberg P, Koch G, Cohen KL. Aqueous vascular endothelial growth factor as a predictor of macular thickening following cataract surgery in patients with diabetes mellitus. Am J Ophthalmol. 2009 Dec;148(6):895-901.e1. doi: 10.1016/j.ajo.2009.07.014. Epub 2009 Oct 17. PMID 19837384
- [Background] Ferguson VM, Spalton DJ. Continued breakdown of the blood aqueous barrier following cataract surgery. Br J Ophthalmol. 1992 Aug;76(8):453-6. doi: 10.1136/bjo.76.8.453. PMID 1390524
- [Background] Dong N, Xu B, Wang B, Chu L, Tang X. Aqueous cytokines as predictors of macular edema in patients with diabetes following uncomplicated phacoemulsification cataract surgery. Biomed Res Int. 2015;2015:126984. doi: 10.1155/2015/126984. Epub 2015 Feb 25. PMID 25811020
- [Background] Patel JI, Hykin PG, Cree IA. Diabetic cataract removal: postoperative progression of maculopathy--growth factor and clinical analysis. Br J Ophthalmol. 2006 Jun;90(6):697-701. doi: 10.1136/bjo.2005.087403. Epub 2006 Mar 15. PMID 16540489